CLINICAL TRIAL: NCT05943678
Title: Novel Metabolic Muscular Biomarkers in Pompe Disease - a Non-invasive
Brief Title: Novel Metabolic Muscular Biomarkers in Pompe Disease - a Non-invasive Magnetic Resonance Exploratory Pilot Study.
Acronym: POMPE
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Scherer, Assoc.Prof. PD Dr., Medical University of Vienna
Other Study IDs: 1868/2022
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pompe Disease; McArdle Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II; Glycogen Storage Disease Type V

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy controls: negative controls
  Interventions: Device: Siemens Magnetom 7T Plus
- Pompe Disease patients
  Interventions: Device: Siemens Magnetom 7T Plus
- McArdle Disease patients: positiv controls
  Interventions: Device: Siemens Magnetom 7T Plus

INTERVENTIONS:
Device: Siemens Magnetom 7T Plus — Magnetic Resonance Spectroscopy

SUMMARY:
Previous studies have indicated that 13C-MRS in the ultra-high 7T magnetic resonance (MR) field is a potential non-invasive measurement method for assessing changes in muscle glycogen levels in PoD patients. However, in a single study, increases in glycogen intermediates were observed using the even more sensitive 31P-MRS technique in a mouse model of PoD and in glycogen storage disease III in humans. In fact, glycolytic intermediates such as phosphomonoesters (PME), measured by phosphorus-31P-MRS in PoD mouse models, were superior to 13C-MRS in monitoring disease progression and quantifying glycogen, indicating a significant clinical potential of 31P-MRS in humans. It has been shown that 31P-MRS can reliably quantify age- and weight-related differences as well as changes in thyroid function in human muscle metabolism. This study conducted by our institute demonstrates that the technique possesses the necessary sensitivity to measure these subtle muscular metabolic changes. However, there are currently no human 31P-MRS muscle data available for PoD. Therefore, we propose a proof-of-principle study to address this knowledge gap and contribute to establishing a new sensitive muscular biomarker that quantifies the primary disease mechanism, namely glycogen formation, for future longitudinal studies on PoD.

ELIGIBILITY:
Inclusion criteria

Patients with PoD and McArdle disease:

* age between 18-70
* Confirmed diagnosis: enzyme activity and/or genetic testing
* body weight > 40kg at screening
* 6-minute walking distance > 75m at screening (only PoD patients)
* Sitting FCV ≥ 30% predicted (only PoD patients)
* "Informed Consent" issued orally and in writing

Healthy volunteers (controls):

• age between 18-70

Exclusion criteria

Patients with PoD and McArdle disease:

* pregnancy (will be assessed prior to MRS measurements using a rapid pregnancy test)
* Involvement of the respiratory musculature
* claustrophobia
* active participation in another clinical trial
* metal devices or other magnetic material in or on the subjects body which will be hazardous for NMR investigation [heart pacemaker, coronary stents and heart valves (in case these devices are not compatible with a 7T MRI), brain (aneurysm) clip, nerve stimulators, electrodes, ear implants, penile implants, colored contact lenses, patch to deliver medications through the skin, coiled spring intrauterine device, vascular filter for blood clots, orthodontic braces, shunt-spinal or ventricular, any metal implants (rods, joints, plates, pins, screws, nails, or clips), embolization coil, or any metal fragments or shrapnel in the body.

Healthy volunteers (controls):

* any known endocrine, metabolic or neurological disorder
* special diets especially ketogenic or atkins diet
* creatine supplementation
* pregnancy (will be assessed prior to MRS measurements using a rapid pregnancy test)
* claustrophobia
* active participation in another clinical trial
* metal devices or other magnetic material in or on the subjects body which will be hazardous for NMR investigation [heart pacemaker, coronary stents and heart valves (in case these devices are not compatible with a 7T MRI), brain (aneurysm) clip, nerve stimulators, electrodes, ear implants, penile implants, colored contact lenses, patch to deliver medications through the skin, coiled spring intrauterine device, vascular filter for blood clots, orthodontic braces, shunt-spinal or ventricular, any metal implants (rods, joints, plates, pins, screws, nails, or clips), embolization coil, or any metal fragments or shrapnel in the body.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with Pompe or McArdle Disease based on enzyme activity and/or genetic testing
  Healthy individuals will serve as controls
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2028-08-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
muscle glycogen concentration | 12 months

SECONDARY OUTCOMES:
muscle phospho-mono-ester concentration (PME) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wary C, Laforet P, Eymard B, Fardeau M, Leroy-Willig A, Bassez G, Leroy JP, Caillaud C, Poenaru L, Carlier PG. Evaluation of muscle glycogen content by 13C NMR spectroscopy in adult-onset acid maltase deficiency. Neuromuscul Disord. 2003 Sep;13(7-8):545-53. doi: 10.1016/s0960-8966(03)00069-5. PMID 12921791
- [Background] Taylor KM, Meyers E, Phipps M, Kishnani PS, Cheng SH, Scheule RK, Moreland RJ. Dysregulation of multiple facets of glycogen metabolism in a murine model of Pompe disease. PLoS One. 2013;8(2):e56181. doi: 10.1371/journal.pone.0056181. Epub 2013 Feb 14. PMID 23457523
- [Background] Baligand C, Todd AG, Lee-McMullen B, Vohra RS, Byrne BJ, Falk DJ, Walter GA. 13C/31P MRS Metabolic Biomarkers of Disease Progression and Response to AAV Delivery of hGAA in a Mouse Model of Pompe Disease. Mol Ther Methods Clin Dev. 2017 Sep 8;7:42-49. doi: 10.1016/j.omtm.2017.09.002. eCollection 2017 Dec 15. PMID 29018835
- [Background] Beiglbock H, Wolf P, Pfleger L, Caliskan B, Fellinger P, Zettinig G, Anderwald CH, Kenner L, Trattnig S, Kautzky-Willer A, Krssak M, Krebs M. Effects of Thyroid Function on Phosphodiester Concentrations in Skeletal Muscle and Liver: An In Vivo NMRS Study. J Clin Endocrinol Metab. 2020 Dec 1;105(12):dgaa663. doi: 10.1210/clinem/dgaa663. PMID 32944774